CLINICAL TRIAL: NCT02932072
Title: Field Evaluation of a Device for Automated Malaria Microscopy (Autoscope Version 2)
Acronym: Autoscope
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: WWARN1602
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2019-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection from finger-prick (maximum 150-200 µL), which will be used to prepare slides.
Oversight: Data Monitoring Committee: No

SUMMARY:
Microscopy remains a key indicator in drug efficacy testing performed in the context of clinical trials for monitoring existing antimalarials or in the context of regulatory clinical trials for registration of new drugs. It is one of the main diagnostic methods for malaria diagnosis in general, as in an ideal setting it can provide low-cost accurate diagnosis, determine the density of parasites in the blood, and accurately differentiate between different malaria parasite species, characteristics vital to the implementation of global plans for drug efficacy monitoring. Malaria rapid tests (RDTs), while useful for case management, do not provide information on the parasite density nor the species differentiation necessary for research and drug efficacy assessment. Microscopy therefore retains key advantages over a number of newer technologies, but its reliability is severely impeded by dependence on high technical competence of the human operators as well as availability of high quality equipment and reagents. Recent studies have demonstrated the frequent poor specificity and sensitivity associated with manual microscopy diagnostics in operational conditions , , . Advances in digital microscopy performance and affordability have now opened the door to potentially significant improvements in the performance of malaria diagnostic microscopy, overcoming serious deficiencies in current drug efficacy assessment, and more broadly in malaria diagnosis and management.

Intellectual Ventures Laboratory (IVL), in collaboration with Global Good Fund (GG), has developed an initial microscope prototype to support its research into dark field imaging of unstained malaria slides. The system consists of low cost electromechanical components for scanning a standard slide, an optical train with a high numerical aperture objective, and an image capture system. Captured images are analyzed with custom image analysis software developed at GG/IVL, using algorithms that are designed for automatic malaria diagnosis, without user input. Additionally, image processing algorithms have been built around detection of Giemsa-stained malaria slides which is the current standard for malaria microscopy. Initial results show excellent potential for sensitivity and specificity which exceeds that of typical manual microscopists in the field. Based on the positive market and needs assessment in January, 2013, given by stakeholders in the malaria diagnostics community, GG/IVL are pursuing improvement and integration of this algorithm into a portable microscope platform with characteristics similar to the prototype microscope already developed at GG/IVL for dark field imaging. The prototype Autoscope was first tested in field settings in Thailand in Nov 2014 - Jan 2015 at clinics operated by the Shoklo Malaria Research Unit (SMRU). The goal of the first field evaluation was to assess the Autoscope in with respect to its diagnostic performance and also its suitability for harsh conditions typically encountered in field clinics. Further, user feedback on the design and functionality was sought. The Autoscope and the accompanying image analysis algorithms have since been further developed and a new version is now available for testing.

DETAILED DESCRIPTION:
Study Design & Procedure The primary purpose of this evaluation is to quantify the diagnostic performance of the Autoscope version 2 prototype in a field setting. The performance of the Autoscope version 2 prototype will be assessed by scanning of negative and positive slides with the Autoscope version 2 and comparing the results with expert microscopy. Plasmodium genus- and species-specific PCR will also be performed as an additional confirmatory test for the detection of malaria parasites and their species if present. Testing by microscopy and Autoscope will be performed in field clinic settings on Giemsa-stained stained slides prepared from febrile patient blood collected from a finger-prick. Patient recruitment will aim to recruit up to 80 slide-confirmed malaria cases (P. falciparum, P. vivax or other species) per country (i.e., total 160 cases) have been included in the study.

Patient procedures Patients who present at the clinic will be screened to assess eligibility. A consent form in the local languages (Karen or Burmese at SMRU sites, Bahasa in South Sumatera at EOCRU site) will be administered to patients with a description of the intentions of this study in order to protect human subjects before any study specific procedures are conducted. It will be clearly stated that participation is voluntary and that the subject or guardian is free to discontinue participation or withdraw consent to participate at any time for any reason without prejudice to future care, and with no obligation to give the reason for discontinuation nor for withdrawal. The subject or guardian will be allowed as much time as needed to consider the information and the opportunity to question the authorized research member, or other independent parties to decide whether they will (or allow his/her charge to) participate in the study. Written informed consent will then be obtained by means of subject or guardian dated signature or thumb print (if unable to write), with signed and dated signature of a witness and dated signature of the person who presented and obtained the informed consent. All individual written informed consent forms will be stored securely.

Children capable of understanding the study (approximately 7 years of age or above for SMRU sites and 12 years of age or above for EOCRU sites) will be asked to sign an assent form. A copy of the signed informed consent document(s) will be given to the participants.

Once informed consent has been obtained, the subject number will be assigned and recorded on the screening and enrollment log. A few drops of blood (maximum of 150-200 µL) will be obtained from a finger-prick and study-specific laboratory procedures as described below will be performed. The patient will then receive clinical care as appropriate according to the routine procedures.

Laboratory procedures All laboratory procedures will be performed according to the applicable standard operating procedures.

At the clinics (Wang Pha, Mawker Tai, Thailand and Hanura, South Sumatera, Indonesia)

* Blood collection from finger-prick (maximum 150-200 µL), which will be used to prepare slides.
* Perform malaria RDT (part of routine practice for malaria detection), prepare 2 slides each with thick and thin blood films, store remainder of blood sample for PCR to detect and determine species of malaria parasites
* Microscopy of Giemsa-stained blood films (microscopists will remain blinded to RDT and Autoscope results), record results
* Run Autoscope detection, record results, store images captured by the device At SMRU and EOCRU
* Review of all slides by expert microscopists (microscopists will remain blinded to RDT and Autoscope results)
* PCR to detect and determine species of malaria parasites At the WWARN Laboratory, Bangkok
* Review of field data to identify discrepant readings and tie-breaker readings in case of discordance between results obtained on site and on re-checking of the slides Quality Assurance
* Quality control performed by WWARN expert microscopists on 20% randomly selected slides or 25 positive and 25 negative slides per country, whichever is greater

The funder is Intellectual Ventures Lab/ Global Good and grant reference PA No.3.

Summary of Results

The sensitivity and specificity of the Autoscope version 2 prototype were 92.2% and 89.2%, respectively. The accuracy was 90.03%. Parasite species were correctly determined in 132/158 slides (83.5%) and kappa value for species detection was 0.60(0.45-0.73). 45.6% of the parasite density estimates from the Autoscope were within 25% range of the reference results, yielding the interclass correlation coefficient (ICC) of 0.78 (95%CI: 0.70-0.83). Bland-Altman plot showed no systematic bias of the measurement. Differences between the 2 counts increased in higher parasite density (correlation coefficient (r) = 0.861, P < 0.001).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age ≥ 6 months to 75 years
* Febrile at presentation or reported within the last 48 hours (>37.5 ºC) and no other obvious diagnosis cause for fever, warranting malaria investigation under routine clinical practice.
* Individual informed assent/consent obtained

Exclusion Criteria:

* Signs of severe malaria as defined by WHO

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eighty slide-confirmed malaria cases (P. falciparum, P. vivax) will be recruited in the study per study site. Accordingly,
  * At EOCRU, with an estimated malaria prevalence of 30% in febrile patients, up to 270 patients will be recruited
  * At SMRU, with an estimated malaria prevalence of 10% in febrile patients, up to 800 patients will be recruited I.e., a total of 1070 subjects with up to 160 malaria positive cases across study sites.
Sampling Method: Probability Sample
Enrollment: 793 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity for malaria parasite detection | 6 months
Diagnostic specificity for malaria parasite detection | 6 months

SECONDARY OUTCOMES:
kappa statistic for parasite species detection | 6 months
Bland-Altman plots for parasite density estimation | 6 months

IPD SHARING:
Plan to Share IPD: No